CLINICAL TRIAL: NCT01270282
Title: Comparison of Single Versus Repeat Doses of AM-101 in the Treatment of Acute Inner Ear Tinnitus
Acronym: TACTT1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Auris Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AM-101-CL-10-02; AM-101-CL-10-02 (Other: Auris Medical)
Record Dates: First submitted 2010-12-30; First posted 2011-01-05 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — PDCD5 protein, rat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- AM-101 0.81 mg/mL (Experimental): Gel for injection; single or triple injection
  Interventions: Drug: AM-101 0.81 mg/mL
- Placebo (Placebo Comparator): Gel for injection; single or triple injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AM-101 0.81 mg/mL
  Arms: AM-101 0.81 mg/mL
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the therapeutic benefit and safety of intratympanic AM-101 injections in comparison to placebo in the treatment of persistent acute inner ear tinnitus.

ELIGIBILITY:
Inclusion Criteria:

* Tinnitus following acute acoustic trauma, acute otitis media, middle ear surgery or inner ear barotrauma; with onset less than three months ago.

Exclusion Criteria:

* Tinnitus that is not completely maskable
* Fluctuating tinnitus
* Intermittent tinnitus
* Meniere's Disease
* Ongoing acute or chronic otitis media or otitis externa.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The change in tinnitus loudness by magnitude estimation from Baseline to 90 days following the last injection | 90 or 104 days

SECONDARY OUTCOMES:
Standard audiological evaluations | 90 or 104 days
  Pure tone audiometry, tympanometry, otoscopy, tinnitus loudness match
Questionnaires evaluating the impact of tinnitus | 90 or 104 days
  Patient global impression of change scale, subjective tinnitus annoyance and loudness, tinnitus handicap questionaire
Pharmacokinetic measures | 3 or 14 days

CONTACTS AND LOCATIONS:
Locations (16):
- United States (5):
  - University of Florida College of Medicine, Gainsville, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Advanced ENT & Allergy, Louisville, Kentucky
  - Summit Medical Group, Berkeley Heights, New Jersey
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
- Belgium (3):
  - UZ Antwerp, Department of ENT, Edegem
  - Gent University Hospital, Department of ENT, Ghent
  - Virga Jesseziekenhuis Hasselt, Hasselt
- Germany (5):
  - HNO Praxis im Schlosscarree, Braunschweig
  - HNO Praxis, Cologne
  - Klinik für Hals-Nasen-Ohrenheilkunde, Kopf- und Halschirurgie, Frankfurt am Main
  - HNO Gemeinschaftspraxis, Heidelberg
  - Bundeswehrkrankenhaus Ulm, Ulm
- Poland (3):
  - NZOZ Laryngologii Wojewodzki Szpital Specjalistyczny, Rzeszów
  - NZOZ Centrum Medyczne LiMED, Tarnowskie Góry
  - Samodzielny Publiczny Centralny Szpital Kliniczny w Warszawie, Warsaw